CLINICAL TRIAL: NCT03460691
Title: Investigation of the Effect of Bariatric Surgery on Knee Pain, Disability, Quality of Life and Central Sensitization
Brief Title: The Effect of Bariatric Surgery to Central Sensitization
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Dr. Burcu Metin Ökmen, Principal Investigator, Bursa Yuksek Ihtisas Training and Research Hospital
Other Study IDs: 2011-KAEK-2017-19/20
Record Dates: First submitted 2018-03-02; First posted 2018-03-09 (Actual); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: Bariatric Surgery; Central Sensitization
Keywords: bariatric surgery; central sensitization; knee pain; function; quality of life
MeSH Terms: interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Group 1:patients who will undergo the bariatric surgery
  Interventions: Procedure: Bariatric surgery

INTERVENTIONS:
Procedure: Bariatric surgery — Bariatric surgery will done to the patients who were morbid obesity

SUMMARY:
Nowadays obesity is emerging as a very common health problem. It has been shown in various studies that obesity may be an important risk factor for the onset and progression of knee osteoarthritis (OA). The aim of this study is to determine the effects of bariatric surgery on knee pain, loss of function, quality of life and central sensitization.

DETAILED DESCRIPTION:
Weight loss in patients with knee OA reduces pain and provides functional improvement. It has been shown that bariatric surgery combined with diet and exercise changes have positive effects on weight loss, knee pain and function.

Neuropathic pain is a disease that affects the somatosensory system or pain that results in a lesion. It has been reported that neuropathic pain is more frequently seen in patients with high body mass index.

The hyperreactivity of the central nervous system (CNS) plays an important role in the chronic pain of OA patients. It has been shown that CNS becomes hypersensitive in people with chronic OA pain and central sensitization phenomenon plays an important role in pain complaints reported by these patients.

The aim of this study is to determine the effects of bariatric surgery on knee pain, loss of function, quality of life and central sensitization.

ELIGIBILITY:
Inclusion Criteria:

* Patients decided to undergo bariatric surgery
* Patients with knee pain more than 3 months.

Exclusion Criteria:

* Patients with mental impairment,
* Patients with inflammatory rheumatic disease,
* Patients who had previously undergone knee surgery

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are morbid obesity and had decided to undergo bariatric surgery
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-03-09 (Estimated); Primary Completion 2018-12-09 (Estimated); Study Completion 2018-12-09 (Estimated)

PRIMARY OUTCOMES:
numeric rating scale (NRS) | 6 months
  It is commonly used to measure the severity of the patients' pain. It consists of a line 10 cm. long and marked with numbers from 0 to 10. The patient is asked to mark the point corresponding to the severity of the pain on this line in the range from 0 (no pain) to 10 (most severe pain).
Western Ontario and McMaster Universities Osteoarthritis Index(WOMAC) | 6 months
  for function
Nottingham Health Profile | 6 months
  for quality of life
Central Sensitization Inventory (CSI) | 6 months
  for central sensitization

CONTACTS AND LOCATIONS:
Overall Officials: Burcu Metin Ökmen, Principal Investigator — Bursa Yuksek Ihtisas Training and Research Hospital